CLINICAL TRIAL: NCT06276101
Title: Phase I Safety and Tolerability Study of NWRD08 in HPV-16 and/or HPV-18 Related Cervical High-grade Squamous Intraepithelial Lesion (HSIL) Patients
Brief Title: NWRD08 DNA Plasmid for HPV-16 and/or HPV-18 Related Cervical HSIL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Newish Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NEWISH-HPV-101
Record Dates: First submitted 2024-02-18; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: High-grade Squamous Intraepithelial Lesion (HSIL)
Keywords: NWRD08; DNA Vaccine; HPV16; HPV18; HSIL
MeSH Terms: conditions — Squamous Intraepithelial Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NWRD08 administered by electroporation (Experimental): Patients will be assigned to three dose groups:1mg, 4mg, and 8mg. Each patient will be administered NWRD08 by electroporation in entire study period. The Maximum Tolerated Dose of NWRD08 will be determined by the classical 3+3 dose escalation schedule. The number of patients will be ranged from 9 to 18.
  Interventions: Biological: NWRD08 administered by electroporation

INTERVENTIONS:
Biological: NWRD08 administered by electroporation — DNA plasmid delivered via IM injection + electroporation using TERESA device

SUMMARY:
This is a single-arm, open label, multi-center Phase 1 clinical study to evaluate the safety and tolerability of HPV-16 and HPV-18-targeted DNA plasmid vaccine (NWRD08) in patients HPV-16 and/or HPV-18 related cervical HSIL.

DETAILED DESCRIPTION:
This study is divided into three dose groups:1mg, 4mg, and 8mg. Each patient will be administered NWRD08 by electroporation in entire study period. The Maximum Tolerated Dose of NWRD08 will be determined by the classical 3+3 dose escalation schedule. The number of patients will be ranged from 9 to 18.

After the completion of treatment, the subjects shall continue to receive safety follow-up until 28 days after the last administration. Colposcopy and biopsy were performed at week 12, if HSIL was identified, loop electro-surgical excisional procedure (LEEP) or cold Knife conization (CKC) will be performed when necessary. The subjects were then followed up at week 36 and all adverse events shall revert to level I or all adverse events shall be clinically stable (whichever is later achieved).

ELIGIBILITY:
Inclusion Criteria:

1. Female aged between 18 and 60 years;
2. histopathological examination/biopsy confirmed HPV-16 and/or HPV-18-associated cervical High-grade squamous intraepithelial lesion (HSIL);
3. The electrocardiograms deemed normal or with abnormalities not considered clinically significant by the site investigators.
4. Major organ functions were normal within 1 week before the first NWRD08 administration: 1) Blood routine: Hemoglobin (Hb) ≥100 g/L; Platelet count (PLT) ≥75×109/L; 2) The liver: Total bilirubin (TB) ≤1.5× upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; Plasma albumin ≥30 g/L; 3)Kidney: Serum creatinine (Scr) ≤1.5×ULN, or creatinine clearance ≥40 mL/min (serum creatinine > 1.5 x ULN);
5. Within 1 week before the first NWRD08 administration, women of childbearing age must have a negative serum pregnancy test and consent to use effective contraception form the signing of the ICF to the end of the study.
6. Have fully understood the study and voluntarily signed the ICF, have good communication with the investigator, and are able to complete all treatments, examinations, and visits stipulated in the study protocol.

Exclusion Criteria:

1. Microscopic or gross evidence of adenocarcinoma-in-situ (AIS), high grade vulvar, vaginal, or anal intraepithelial neoplasia or invasive cancer in any histopathologic specimen at screening;
2. Pregnant, breastfeeding or considering becoming pregnant during the study;
3. Administration of any non-live vaccines within 2 weeks prior to the first NWRD08 administration;
4. Administration of any live vaccines within 4 weeks prior to the first NWRD08 administration;
5. Treatment for cervical HSIL within 4 weeks prior to the first NWRD08 administration;
6. Any metallic implants/implanted electric devices around the intended sites of electroporation (deltoid muscles);
7. Participated in another clinical trial or was under observation in another clinical trial within 30 days prior to screening;
8. Continuous (more than 1 week) glucocorticoid therapy (dose equivalent to prednisone > 10 mg/ day) within 30 days prior to screening, except hormone replacement therapy, intratracheal, ocular and topical administration;
9. A history of immune deficiency or autoimmune diseases (e.g., rheumatoid joint disease, systemic lupus erythematosus, multiple sclerosis, etc.);
10. Current or intended use of disease-modifying antirheumatic drugs (e.g., azathioprine, cyclophosphamide, cyclosporin and methotrexate) and biologic drugs (e.g., infliximab, adalimumab and etanercept);
11. Continuous (more than 1 week) use of immunosuppressive agents. (e.g., cyclosporin, tacrolimus, azathioprine, 6-mercaptoputine and antilymphocyte globulin, etc.);
12. Patients with a history of solid organ or bone marrow transplantation;
13. With uncontrolled severe infection (> grade 2 NCI-CTCAE adverse events, version 5.0);
14. Patients with a history of human immunodeficiency virus (HIV) infection or carriers of syphilis;
15. Patients who are found to have active zoster virus infections;
16. Patients with serious other organ dysfunction or cardiopulmonary diseases;
17. Epilepsy that requires treatment with medication (e.g. steroids or antiepileptic drugs);
18. Had or currently has other malignancies (with the exception of adequately treated and completely cured ductal carcinoma in situ of the breast, carcinoma in situ of the cervix, basal cell carcinoma of the skin, superficial bladder tumor, or any malignancy that was cured more than 5 years before study entry);
19. A known history of albumin allergy, or severe allergy, or allergic disease, or allergic constitution, or severe iodine contrast allergy, meeting any of these criteria;
20. Patients with clinically significant heart disease or medical history;
21. Severe mental illness;
22. A history of drug or alcohol abuse;
23. Pregnant or lactating women, or women of childbearing age with positive blood pregnancy tests, or women of reproductive age and their spousal not willing to use contraception during and up to 6 months following completion of the study;
24. Patients deemed by the investigator to be ineligible for this clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Safety | From first administration of NWRD08 to 24 weeks (Week36) after the last administration.
  All adverse events (AE) will be determined based on the rate and severity grade of events, including incidence and severity of serious adverse events (SAE) (according to NCI-CTCAE Standard version 5.0 of common Terms for Adverse Events). The grade of injection-site AEs will be determined on the basis of the Guidelines for Adverse Event Classification Standards for Clinical Trials of Preventive Vaccines (2019) issued by the National Medical Products Administration.
Dose-limiting toxicity (DLT) | From first administration of NWRD08 to 28 days after the last administration
  t would be determined based on the rate and severity grade of events or abnormalities through evaluating systemic or local adverse events, clinical laboratory test results, vital signs that is definitely, probably, or possibly related to the test drug occurring within 28 days of the last dosing will be classified as DLT during dosing climb.

SECONDARY OUTCOMES:
Immunogenicity | At week 0, week 2, week 4, week 6, week 8, week 10, week 12 and week 36.
  Immunologic reactogenicity by measuring HPV16/18 E6/E7 specific T cell response (IFN-γ ELISPOT) and anti-HPV16/18 E6/E7antibodies (ELISA) in blood samples.
Histopathology outcome and HPV Viral clearance | Week 12
  Number of subjects with virologically-proven clearance of HPV 16 or 18 and number of subjects with histopathological regression of cervical lesions to CIN 1 or normal.
The recommended phase II dose (RP2D) | Week 12
  The recommended phase II dose (RP2D) was selected on the basis of tolerability during the safety expansion.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiang, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication
Access Criteria: by publication